CLINICAL TRIAL: NCT00045396
Title: A Phase II Study of the Farnesyltransferase Inhibitor ZARNESTRA (Tipifarnib, R115777, NSC #702818, IND #58,359) in Complete Remission Following Induction and/or Consolidation Chemotherapy in Adults With Poor-Risk Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplasia (MDS).
Brief Title: A Phase II Study Of The Farnesyltransferase Inhibitor ZANESTRA (R115777, NSC #702818, IND #58,359) In Complete Remission Following Induction And/Or Consolidation Chemotherapy In Adults With Poor-Risk Acute Myelogenous Leukemia (AML) And High-Risk Myelodysplasia (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03158; J0252; U01CA070095 (NIH); U01CA069854 (NIH)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); de Novo Myelodysplastic Syndromes; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities | interventions — tipifarnib

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive oral tipifarnib twice daily on days 1-14. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra

SUMMARY:
Tipifarnib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Phase II trial to study the effectiveness of tipifarnib in treating patients who have acute myeloid leukemia or myelodysplastic syndrome in first complete remission

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the duration of disease-free survival (DFS) and overall survival (OS) when ZARNESTRA is administered after intensive induction and consolidation chemotherapy to adults with poor risk acute myelogenous leukemia (AML) or high-risk myelodysplasia (MDS) in first complete remission (CR).

SECONDARY OBJECTIVES:

I. To determine the tolerability and toxicities of ZARNESTRA when administered in a chronic dosing schedule over a 48 week period to adults in first CR following intensive cytotoxic chemotherapies.

OUTLINE: This is a multicenter study.

Patients receive oral tipifarnib twice daily on days 1-14. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 14-44 patients will be accrued for this study within 11-15 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathological Confirmation of the Diagnosis of AML, MDS
* PMNs >= 1,000/ul
* Platelets >= 30,000/ul
* Hematocrit >= 27% and/or Hemoglobin >= 9 gm/dl unsupported
* ECOG Performance Status 0-2
* Patients must be able to give informed consent
* Female patients of childbearing age must have negative pregnancy test
* AST, ALT and Alkaline Phosphatase =<2.5 x normal
* Bilirubin =< 1.5 x normal
* Serum Creatinine =< 2.0 mg/dl or Creatinine Clearance >= 40 ml/min
* Left Ventricular Ejection Fraction >= 25%
* Patients with poor-risk AML or high-risk MDS who have completed both induction and consolidation chemotherapy; poor risk AML is defined by one or more of the following characteristics:

  * Antecedent Hematologic Disorder
  * AML Arising from MDS
  * Therapy-related AML
  * Age >= 60 (in absence of favorable cytogenetics)
  * Adverse Cytogenetics (i.e., -5/5q, -7/7q, +8, 20q-, 11q23 abnormalities, complex karyotype; other abnormalities may be considered at discression of study chair)
  * Hyperleukocytosis at diagnosis (Blasts >= 30,000/mm^3 at diagnosis in absence of favorable cytogenetics)

High Risk MDS is defined by one or more of the following characteristics:

* RAEB and RAEB-t, with IPSS Score >= 1.5 (adverse cytogenetics, > 10% marrow blasts, cytopenias in at least 2 lineages): See Appendix E (Greenberg, et al. Blood 89:2079-2088,1997)36
* CMML with > 5% marrow blasts
* Therapy-related MDS

Exclusion Criteria:

* Any previous treatment with ZARNESTRA
* Ongoing participation in any Phase II or III clinical trial where DFS and OS are primary endpoints (unless patient is withdrawn from that trial)
* Acute promyelocytic (FAB M3) subtype
* Presence of (8;21) translocation or inversion 16 genotype as sole abnormality
* Eligible for curative allogeneic stem cell transplantation
* Known allergy to imidazole drugs (e.g., ketoconazole, miconazole)
* Presence of Residual AML (> 5% marrow blasts) or MDS, as Determined by Morphology, Flow Cytometry, and/or Cytogenetics
* Active, Uncontrolled Infection
* Disseminated Intravascular Coagulation
* Active CNS Leukemia
* Concomitant Chemotherapy, Radiation Therapy or Immunotherapy
* Women who are pregnant or lactating will not be eligible for this trial, as the investigational agent may be harmful to the developing fetus or nursing infant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2002-06; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 6 months
  The trial is a success if greater than 45% of patients survive to 6 months. Comparing this to the null hypothesis of 25% survival, we have 84% power to detect this difference using an exact 2-sided binominal test of proportions for alpha of 0.10. This assumes no censoring occurs before 6 months.

SECONDARY OUTCOMES:
Tolerability and toxicities of ZARNESTRA when administrated in a chronic dosing schedule over a 48-week period to adults in first CR following intensive cytotoxic chemotherapy | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States